CLINICAL TRIAL: NCT02278159
Title: Evaluation of the Integrated Home Dialysis Model
Status: Completed | Type: Observational
Sponsor: Princess Alexandra Hospital, Brisbane, Australia (Other)
Collaborators: Baxter Healthcare Corporation (Industry)
Responsible Party: Principal Investigator, David Johnson, Director of Metro South and Ipswich Nephrology and Transplant Services (MINTS) Medical Director, Queensland Renal Transplant Services Professor of Medicine (University of Qld), Princess Alexandra Hospital, Brisbane, Australia
Other Study IDs: ANZ41367
Record Dates: First submitted 2014-06-19; First posted 2014-10-29 (Estimated); Last update posted 2014-10-29 (Estimated); Status verified 2014-10

CONDITIONS: Kidney Failure, Chronic
Keywords: end-stage kidney disease; peritoneal dialysis; home hemodialysis; technique survival; patient survival
MeSH Terms: conditions — Kidney Failure, Chronic | interventions — Peritoneal Dialysis; Hemodialysis, Home

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (4):
- Peritoneal dialysis only: Patient on PD modality 90 days after renal replacement therapy initiation and not transferred to HHD
  Interventions: Procedure: Peritoneal dialysis
- Home hemodialysis only: Patient on HHD 90 days after renal replacement therapy initiation and not transferred to PD
  Interventions: Procedure: Home hemodialysis
- PD and HHD: Patient on PD 90 days after RRT initiation and transferred to HHD less than 90 days after PD failure
  Interventions: Procedure: Peritoneal dialysis; Procedure: Home hemodialysis
- HHD and PD: Patient on HHD after RRT initiation and transferred to PD less than 90 days after HHD failure
  Interventions: Procedure: Peritoneal dialysis; Procedure: Home hemodialysis

INTERVENTIONS:
Procedure: Peritoneal dialysis
  Groups: HHD and PD; PD and HHD; Peritoneal dialysis only
Procedure: Home hemodialysis
  Groups: HHD and PD; Home hemodialysis only; PD and HHD

SUMMARY:
The purpose of this study is to evaluate which home dialysis modality pattern (home hemodialysis [HHD], peritoneal dialysis [PD] or a combination of both, e.g. PD and then HHD) allows for the longest home dialysis survival, as defined by the time dialysed in a home environment. The investigators hypothesize that patients transferred from one home modality to another will have a longer home dialysis survival compared to patients treated only with PD or HHD.

ELIGIBILITY:
Inclusion Criteria:

* Patients with PD/HHD 90 days after RRT initiation between January 1, 2000 and December 31, 2012 reported in ANZDATA
* ≥ 18 years

Exclusion Criteria:

* Less than 90 days of dialysis
* < 18 years
* Patients transferred to Australia/New Zealand after initiation of dialysis in another country

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with home dialysis as the first renal replacement therapy [RRT] modality (defined by the dialysis modality at 90 days) in Australia and New Zealand as reported in Australia and New Zealand Dialysis and Transplant Registry [ANZDATA]
Sampling Method: Non-Probability Sample
Enrollment: 11600 (Actual)
Dates: Start 2000-01; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Home dialysis survival | Survival analysis; specific analysis at 5 years after dialysis initiation
  Time to first patient death or home dialysis technique failure for each home dialysis modalities, censored for transplantation and loss to follow-up

SECONDARY OUTCOMES:
Patient survival, censored for technique failure | Survival analysis, specific analysis at 1,2 5 years after dialysis initiation
  Patient survival on each specific home dialysis modality, censored for technique failure, transplantation and loss to follow-up
Home technique survival, censored for death | survival analysis, specific analysis at 1,2 5 years after dialysis initiation
  Home dialysis technique survival for each home dialysis modality, censored for patient death, transplantation and loss to follow-up

OTHER OUTCOMES:
Home dialysis survival, case-control analysis | survival analysis, specific analysis at 1,2 5 years after dialysis initiation
  Case-control analysis will be performed in order to address immortal bias in patients classified in the "switching"categories (PD-HHD or HHD-PD). Since we expect the HHD-PD group to be small, this analysis will be performed only with the 3 other groups (PD-HHD, PD only and HHD only). Patients treated successively with PD and HHD (cases) will be matched (by age and diabetes status) to patient treated with PD only and HHD only (controls).